CLINICAL TRIAL: NCT00534976
Title: A Double-Blind, Placebo-Controlled, Multicenter, Crossover Study to Evaluate the Effects of a Single Oral Dose of Montelukast, Compared With Placebo, on Exercise-Induced Bronchoconstriction (EIB) in Pediatric Patients Aged 4 to 14 Years
Brief Title: The Effect of Montelukast on Difficulty in Breathing After Exercise in Pediatric Patients (MK0476-377)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-377; 2007_586
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2022-01

CONDITIONS: Exercise-induced Bronchoconstriction (EIB)

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Montelukast Sodium (Experimental): Participants 4-5 years: A single dose of 4 mg Montelukast chewable tablet daily, crossing over to matching placebo (Pbo) after a 3- to 7-day washout period (no participants 4-5 years were enrolled)
  Participants 6-14 years: A single dose of 5 mg Montelukast chewable tablet daily, crossing over to matching Pbo after a 3- to 7-day washout period
  Interventions: Drug: Comparator: montelukast sodium
- Placebo (Experimental): Participants 4-5 years: A single dose of 4 mg Pbo chewable tablet daily, crossing over to Montelukast 4 mg chewable tablet after a 3- to 7-day washout period (no participants 4-5 years of age were enrolled)
  Participants 6-14 years: A single dose of 5 mg Pbo chewable tablet daily, crossing over to Montelukast 5 mg chewable tablet after a 3- to 7-day washout period
  Interventions: Drug: Comparator: Comparator: placebo (unspecified)

INTERVENTIONS:
Drug: Comparator: montelukast sodium — Patients 4-5 years: 4 mg Montelukast chewable tablet daily
  Patients 6-14 years: 5 mg chewable tablet daily
  Arms: Montelukast Sodium
Drug: Comparator: Comparator: placebo (unspecified) — Patients 4-5 years: 4 mg Pbo chewable tablet daily
  Patients 6-14 years: 5 mg Pbo chewable tablet daily
  Arms: Placebo

SUMMARY:
This study will see if there is a change in breathing after exercising when the child receives study drug ( montelukast or placebo). Breathing will be measured by a spirometer before exercising and measured again several times after exercising.

ELIGIBILITY:
Inclusion Criteria:

* The child is 4 years to 14 years of age
* The child is a non smoker
* The child has exercise-induced bronchoconstriction (EIB)

Exclusion Criteria:

* The child has active or chronic breathing disease, other than asthma
* The child has required insertion of a breathing tube for asthma
* The child had major surgery within the last 4 weeks
* The child is currently in the hospital
* The child has or had an upper respiratory tract infection within the last 2 weeks
* The child has been hospitalized or visited the emergency room or had a change in their medication for asthma within the last 4 weeks
* The child has been in a research study in the last 4 weeks
* The child has stomach, brain, heart, kidney or liver disease
* The child drinks more that 4 caffeinated drinks a day

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 364 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wasfi YS, Kemp JP, Villaran C, Massaad R, Xin W, Smugar SS, Knorr BA, Philip G. Onset and duration of attenuation of exercise-induced bronchoconstriction in children by single-dose of montelukast. Allergy Asthma Proc. 2011 Nov-Dec;32(6):453-9. doi: 10.2500/aap.2011.32.3482. PMID 22221440

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 364 participants screened for inclusion, 298 participants were excluded during screening and were not randomized. The remaining 66 participants met inclusion criteria and were randomly allocated to one of the two treatment sequences.
Groups:
- Montelukast/ Placebo: In Period I (screening period/ placebo run-in) participants received a single-blind dose of matching-image placebo. In Period II, participants 4-5 years of age were randomized to receive one Montelukast 4-mg chewable tablet (single dose). Period III was the crossover to one matching placebo 4-mg chewable tablet (single dose) after a 3- to 7-day washout period. No participants 4-5 years of age were randomized, so the 4-mg doses were not dispensed. Participants 6-14 years of age were randomized to receive one Montelukast 5-mg chewable tablet (single dose) in Period II, crossing over to one matching placebo 5-mg chewable tablet (single dose) in Period III after a 3- to 7-day washout period.
- Placebo/ Montelukast: In Period I (screening period/ placebo run-in) participants received a single-blind dose of matching-image placebo. In Period II, participants 4-5 years of age were randomized to receive one placebo 4-mg chewable tablet (single dose). Period III was the crossover to one Montelukast 4-mg chewable tablet (single dose) after a 3- to 7-day washout period. No participants 4-5 years of age were randomized, so the 4-mg doses were not dispensed. Participants 6-14 years of age were randomized to receive one placebo 5-mg chewable tablet (single dose) in Period II, crossing over to one Montelukast 5-mg chewable tablet (single dose) in Period III after a 3- to 7-day washout period.
Period: Period 1: Placebo Run-in
Arm/Group | Montelukast/ Placebo | Placebo/ Montelukast
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0
Period: Period 2: Treatment Montelukast/ Placebo
Arm/Group | Montelukast/ Placebo | Placebo/ Montelukast
Started | 33 | 33
Completed | 33 | 32
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Period 3: Crossover Placebo/ Montelukast
Arm/Group | Montelukast/ Placebo | Placebo/ Montelukast
Started | 33 | 32
Completed | 31 | 32
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast/ Placebo | Placebo/ Montelukast | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (2.3) | 11.5 (1.8) | 11.2 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Fall in Forced Expiratory Volume in 1 Second (FEV1) After Exercise Challenge at 2 Hours Postdose
Description: Maximum Percent Fall in FEV1 was defined as the % change from pre-exercise baseline FEV1 to the lowest FEV1 within 60 mins (minutes) after exercise. Spirometry measurements were taken 5 mins prior to each exercise challenge and immediately, 5, 10, 15, 30, 45, & 60 mins after each exercise challenge. The 2-hour exercise challenges occurred 2 hours after the witnessed dose of study medication. The calculation used to produce the results was [100*(1-(X/Y))] where X= the lowest FEV1 within 60 mins after exercise & Y= pre-exercise baseline FEV1. Smaller values mean greater response to therapy.
Time Frame: Pre-exercise baseline and 0-60 minutes after the exercise challenge performed 2 hours post-dose
Population: The analysis of efficacy data was carried out using a completers analysis population. This population included all randomized patients who received the witnessed dose of study drug in both active treatment periods and had at least one post-exercise FEV1 measurement in both active treatment periods.
Measure: Mean (Standard Deviation); unit: Percent fall in FEV1
Groups:
- Montelukast: In Period I (screening period/ placebo run-in) participants received a single-blind dose of matching-image placebo. Participants 6-14 years of age were randomized to receive one Montelukast 5-mg chewable tablet (single dose) in Period II or Period III, according to the randomized treatment sequence assigned. Period II and Period III were separated by a washout period of 3-7 days.
- Placebo: In Period I (screening period/ placebo run-in) participants received a single-blind dose of matching-image placebo. Participants 6-14 years of age were randomized to receive one matching placebo 5-mg chewable tablet (single dose) in Period II or Period III, according to the randomized treatment sequence assigned. Period II and Period III were separated by a washout period of 3-7 days.
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 64 | 64
Percent fall in FEV1 | 15.35 (9.47) [12.60 to 18.11] | 20.00 (15.75) [17.25 to 22.76]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.020, ANOVA; Difference in least square means = -4.65 — Montelukast minus placebo

2. Secondary Outcome: Maximum Percent Fall in FEV1 After Exercise Challenge at 24 Hours Post-dose
Description: Maximum Percent Fall in FEV1 was defined as the % change from pre-exercise baseline FEV1 to the lowest FEV1 within 60 mins after exercise. Spirometry measurements were taken 5 mins prior to each exercise challenge and immediately, 5, 10, 15, 30, 45, & 60 mins after each exercise challenge. The 24-hour exercise challenges occurred 20-24 hours after the witnessed dose of study medication. The calculation used to produce the resulted results was [100*(1-(X/Y))] where X= the lowest FEV1 within 60 mins after exercise & Y= pre-exercise baseline FEV1. Smaller values mean greater response to therapy.
Time Frame: Pre-exercise baseline and 0-60 minutes after the exercise challenge performed 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent fall in FEV1
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 62 | 62
percent fall in FEV1 | 12.96 (10.38) [10.81 to 15.04] | 17.22 (12.06) [15.14 to 19.36]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.005, ANOVA; Difference in least square means = -4.33 — Montelukast minus placebo

3. Secondary Outcome: Area Under the Curve for FEV1 Percent Fall From Pre-exercise Baseline to 60 Minutes Following Exercise Challenge (AUC0-60 Min) at 2 Hours Post-dose
Description: AUC0-60min was defined as the Area Under the Curve for FEV1 percent change from pre-exercise baseline to the 60 mins following exercise challenge. The area was computed by applying the trapezoidal rule, and including only the area below the pre-exercise baseline. If a participant received β-agonist during the 60 mins after the exercise challenge, the FEV1 measurements obtained after β-agonist administration were excluded and the last pre-rescue FEV1 measurement was carried forward to the 60 mins time point in the calculation of the AUC0-60 min. Smaller values mean greater response to therapy.
Time Frame: Pre-exercise baseline to 60 minutes after the exercise challenge performed 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent fall * minute
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 64 | 64
percent fall * minute | 294.50 (278.46) [221.73 to 367.27] | 415.37 (375.94) [342.60 to 488.13]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.022, ANOVA; Difference in least square means = -120.86 — Montelukast minus placebo

4. Secondary Outcome: Area Under the Curve for FEV1 Percent Fall From Pre-exercise Baseline to 60 Minutes Following Exercise Challenge (AUC0-60 Min) at 24 Hours Post-dose
Description: as for outcome 3
Time Frame: Pre-exercise baseline to 60 minutes after the exercise challenge performed 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent fall * minute
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 62 | 62
percent fall * minute | 229.19 (233.93) [160.44 to 295.51] | 349.59 (315.29) [283.26 to 418.34]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.013, ANOVA; Difference in least square means = -122.82 — Montelukast minus placebo

5. Secondary Outcome: Time to Recovery From Maximum Percent Fall in FEV1 at 2 Hours Post-dose
Description: This endpoint was defined as the duration between the time at which the maximum percent fall in FEV1 occurred & the time when the percent fall in FEV1 returned to within 5% of the pre-exercise baseline for the first time.
  Spirometry measurements were taken 5 mins prior to each exercise challenge & immediately, 5, 10, 15, 30, 45, & 60 mins after each exercise challenge. If participant had not returned to within 5% of the pre-exercise FEV1 value by 60 mins, then measurements were obtained at 75 & 90 mins.
  The 2-hour exercise challenges occurred 2 hours after the witnessed dose of medication.
Time Frame: 0-60 minutes and 0-90 minutes after the exercise challenge at 2 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 64 | 64
Minutes | 16.21 (22.01) [10.01 to 22.42] | 24.48 (27.91) [18.27 to 30.68]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.064, ANOVA; Difference in least square means = -8.27 — Montelukast minus placebo

6. Secondary Outcome: Time to Recovery From Maximum Percent Fall in FEV1 at 24 Hours Post-dose
Description: This endpoint was defined as the duration between the time at which the maximum percent fall in FEV1 occurred & the time when the percent fall in FEV1 returned to within 5% of the pre-exercise baseline for the first time. Spirometry measurements were taken 5 mins prior to each exercise challenge & immediately, 5, 10, 15, 30, 45 & 60 mins after each exercise challenge. If participant had not returned to within 5% of the pre-exercise FEV1 value by 60 mins, then measurements were obtained at 75 & 90 mins. The 24-hour exercise challenges occurred 20-24 hours after the witnessed dose of medication.
Time Frame: 0-60 minutes and 0-90 minutes after the exercise challenge at 24 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 62 | 62
Minutes | 11.58 (16.51) [6.42 to 16.56] | 18.46 (22.66) [13.48 to 23.62]
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 0.054, ANOVA; Difference in least square means = -7.06 — Montelukast minus Placebo

7. Secondary Outcome: Number of Participants Requiring Rescue Medication at 2 Hours Postdose
Description: This endpoint was defined as the number of participants requiring rescue medication with β-agonist within the 90 mins following exercise challenge. The 2-hour exercise challenges occurred 2 hours after the witnessed dose of study medication.
Time Frame: 0-90 minutes after the exercise challenge at 2 hours postdose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 64 | 64
participants | 1 [-9.27 to 5.63] | 2
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; p = 1.000, McNemar — P-value provided is for comparison between the two proportions: Montelukast versus placebo; Difference in Proportions = -1.6 — Montelukast minus placebo

8. Secondary Outcome: Number of Participants Requiring Rescue Medication at 24 Hours Postdose
Description: This endpoint was defined as the number of participants requiring rescue medication with β-agonist within the 90 mins following exercise challenge. The 24-hour exercise challenges occurred 20-24 hours after the witnessed dose of study medication.
Time Frame: 0-90 minutes after the exercise challenge at 24 hours postdose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 62 | 62
Participants | 0 [-11.02 to 3.06] | 2
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority or Other; Difference in Proportions = -3.2 — Montelukast minus placebo

ADVERSE EVENTS:
Description: The analysis of safety data was carried out using an all patients as treated (APaT) population. This population included all randomized patients who received at least one dose of study treatment.
Arm/Group | Montelukast | Placebo
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/66
Other Adverse Events (participants affected / at risk) | 0/65 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to a multicenter publication, or 24 months after completion of the study, whichever comes first, an investigator may publish the results for their study site independently. However, the SPONSOR does not recommend separate publication of individual study site results. The SPONSOR must have the opportunity to review all proposed communications regarding this study 60 days prior to submission. Any information identified by the SPONSOR as confidential must be deleted.